CLINICAL TRIAL: NCT05750485
Title: Pupilometric Evaluation of Nociception in Patients With Orthopedic Impairment Under Procedural Sedation With Propofol in the Context of the Use of the ALGISCAN Device in the Vital Emergency Department in Pasteur 2 Hospital, Nice France
Brief Title: Pupilometric Evaluation of Patients Under Procedural Sedation With Propofol
Acronym: ALGISAP 2023
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Urgences01_Hamard
Record Dates: First submitted 2023-02-07; First posted 2023-03-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pupilometric evaluation under procedural sedation with propofol
  Interventions: Other: Pupilometric evaluation

INTERVENTIONS:
Other: Pupilometric evaluation — Pupilometric evaluation under procedural sedation with propofol

SUMMARY:
Procedural sedation involves the administration of sedative medications that allow patients to tolerate painful procedures. Procedural sedation has been formally recommended by experts from the French Society of Emergency Medicine (SFMU) since 2010 and procedural sedation using propofol in emergency departments has been recommended by the American College of Emergency Physicians in 2018.

Propofol monotherapy is now widely used in emergency medicine (EM) in France as part of procedural sedation for performing painful procedures, however propofol has no analgesic properties per se .

Pupilometry makes it possible to study the depth of analgesia by evaluating the body's nociceptive response via the ANS by studying the pupil diameter.

This technique would allow the evaluation of the analgesia level in patients sedated by PROPOFOL during the realization of painful procedures. Variations in pupil diameter during painful procedures under procedural sedation in an emergency department will be assesed in this study. Secondly, patients satisfaction following the procedure will also be evaluated by the use of the French version of the "ISAS-F", the Iowa Satisfaction with Anesthesia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* patient admitted at vital emergency room,
* patient with an orthopedic trauma,
* patient under procedural sedation with PROPOFOL.

Exclusion Criteria:

* Patient's refusal of pupilometry measurement.
* Pre-existing pupil abnormalities.
* history of pathologies with dysautonomic impairment (advanced diabetes, systemic amyloidosis, multiple sclerosis, uncontrolled hypertension, ...).
* Recent administration of Metoclopramide, Droperidol, Clonidine, Dexmedetomidine
* Nitrous oxide prior to procedural sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted at vital emergency room, consecutive to an orthopedic trauma, for the performance of a painful procedure under procedural sedation with PROPOFOL.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
pupil dilation reflex | up to 10 minutes
  Amplitude of pupil dilation reflex (PRD, in % change in pupil diameter)

SECONDARY OUTCOMES:
Pupil diameter using the Algiscan device | up to 10 minutes
  Pupil diameter using the Algiscan device during the painful procedure.
Pupil diameter variation using the Algiscan | up to 10 minutes
  Pupil diameter variation using the Algiscan device during the painful procedure.
Heteroevaluation of the patient's maximal pain | up to 10 minutes
  Heteroevaluation of the patient's maximal pain by the doctor, caregiver or nurse using the Algoplus scale (from 0 to 5) during the painful procedure.
Patient's minimal Ramsay score | up to 10 minutes
  Patient's minimal Ramsay score (from 0 to 6) during painful procedure
Level of sedation | up to 10 minutes
  Level of sedation ("qCON" consciousness index)as continuously measured by the Conox® device
Patient satisfaction | up to 10 minutes
  Patient satisfaction as evaluated by the study questionnaire When patients are fully awaked
feasibility of the measurement | up to 10 minutes
  Assessment of the feasibility of the measurement by the personnel who carried out the pupilometry measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No